CLINICAL TRIAL: NCT03155048
Title: The Effects of Transdermal Estradiol and Oral Estradiol Valerate on Clinical Outcomes of Frozen-thawed Embryo Transfer Cycles: A Randomized Clinical Trial
Brief Title: The Effects of Estrogen on Artificial Endometrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sisli Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Prof. Dr. Semra Kahraman, Director of ART and Genetics Center of Memorial Sisli Hospital, Memorial Sisli Hospital, Istanbul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EndometrialpreparingSK002
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Estrogen Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral estradiol group (Active Comparator): patients with the usage of 6 milligrams/day oral estradiol
  Interventions: Drug: oral estrogen replacement therapy
- estradiol transdermal patch group (Active Comparator): patients with the usage of 3.9 milligrams estradiol transdermal patch
  Interventions: Drug: Estradiol transdermal patch

INTERVENTIONS:
Drug: oral estrogen replacement therapy — oral estradiol group for endometrial preparation
  Arms: oral estradiol group
Drug: Estradiol transdermal patch — transdermal estradiol group for endometrial preparation
  Arms: estradiol transdermal patch group

SUMMARY:
In this prospective randomized trial, the parameters of the frozen-thawed embryo transfer (FET) cycles were analyzed. This study was undertaken in the Department of Assisted Reproductive Technologies and Reproductive Genetics Center at Istanbul Memorial Hospital with approval of the local ethics committee. The aim of this prospective randomized clinical trial was to compare two methods of endometrial preparation for FET, oral estradiol and estradiol transdermal patch.

DETAILED DESCRIPTION:
In this prospective randomized trial, the parameters of the frozen-thawed embryo transfer (FET) cycles were analyzed. This study was undertaken in the Department of Assisted Reproductive Technologies and Reproductive Genetics Center at Istanbul Memorial Hospital with approval of the local ethics committee. The aim of this prospective randomized clinical trial was to compare two methods of endometrial preparation for FET, oral estradiol and estradiol transdermal patch.

A total number of 317 patients who underwent frozen -thawed embryo transfer cycles were enrolled in this study and randomized to two groups including 160 patients with the usage of 6 milligrams/day oral estradiol and 154 patients with the usage of 3.9 milligrams estradiol transdermal patch. Randomization was done with http://www.randomization.com. The patients were given sufficient information to provide written informed consent. All the women underwent intracytoplasmic sperm injection (ICSI).

Treatment protocols: All the patients selected for the research were primed for a frozen transfer using two different ways of exogenous steroid therapy.

In the study group with transdermal route (n=154), 3.9 milligrams of estradiol transdermal patch was applied every other day from the second day of menstruation cycle, and each patch was removed after day. In the control group with oral route (n=160), at the time of cycle, 6 milligrams of oral estradiol valerate was started daily. In both groups, clinical monitoring was done by transvaginal ultrasound from the 11th day of the cycle to measure endometrial thickness. If endometrial thickness was more than 7 millimeter, 90 milligrams vaginal natural progesterone was added. Embryo transfer was done after 5 days.

The primary outcome measure was endometrial thickness on the day of progesterone administration. The secondary outcome measures were chemical and clinical pregnancy, implantation rates, abortion rates, live birth rates, and cycle cancellation rate.

ELIGIBILITY:
Inclusion Criteria:

* All the women with at least one day 5 or 6 blastocyst
* Appropriate endometrial thickness is more than 7 millimeters on the 14th day of artificial endometrial preparation cycle
* Age under 38 years
* Follicle stimulating hormone less than 12 IU/Liter
* No more than 2 previous treatment cycles
* No history of recurrent spontaneous abortions

Exclusion Criteria:

* Polycystic ovarian syndrome (> 30 cumulus oocyte complexes retrieved at the pick-up)
* Endocrine or metabolic disorder
* Endometriosis
* Embryos derived from donated gametes
* Any underlying diseases (kidney, liver or heart diseases)
* Bad-quality embryos
* Uterine malformation
* Endometrial polyp
* Severe male factor (Azoospermia)
* Body mass index more than 30
* Thrombophilia

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness on the day of progesterone administration | 6 months
  In frozen thawed embryo transfer cycles, endometrial preparation with estrogen was performed. Estrogen was applied from the second day of menstruation cycle to 11th day of cycle. Endometrial thickness was measured by transvaginal ultrasound. If endometrial thickness was more than 7 millimeters, endometrial thickness was ready for embryo transfer on the day of progesterone administration.

SECONDARY OUTCOMES:
Implantation rate | 12 months
  The effects of transdermal estradiol and oral estradiol valerate on implantation rates were evaluated. Implantation rates are described as gestational sacs seen by transvaginal ultrasound per embryo transfer.

OTHER OUTCOMES:
Clinical Pregnancy rate | 12 months
  The effects of transdermal estradiol and oral estradiol valerate on clinical pregnancy rate were evaluated. Clinical pregnancy rate is measured with a pregnancy where an ultrasound scan has shown at least one fetal heartbeat per embryo transfer.
Live birth rate | 12 months
  The effects of transdermal estradiol and oral estradiol valerate on live birth rate were evaluated. Live birth rate is described as live birth per embryo transfer.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sisli Hospital ART and Genetics Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No